CLINICAL TRIAL: NCT06988163
Title: OACareTools Primary Care-Led Usability & Scalability Pilot Study (OACareTools PLUS)
Brief Title: Osteoarthritis Care Tools for Primary Care Providers
Acronym: OACareTools
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-2284; 1 U48DP006837-01-00 (Other Grant/Funding Number: Centers for Disease Control and Prevention); 1U48DP006837-01 (NIH)
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Arthritis; Osteo Arthritis Knee
Keywords: healthcare providers; arthritis; primary care
MeSH Terms: conditions — Arthritis | interventions — Walking; methyl hydroxyethyl cellulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthcare providers (Experimental): Healthcare providers will receive the intervention, OACareTools+, which involves a training session on, patient resources about, and provider referral to Walk With Ease.
  Interventions: Behavioral: OACareTools+
- Patients (Experimental): A subset of patients who are referred through OACareTools+ by their provider and participate in Walk With Ease will provide feedback on their experience with the referral process to Walk With Ease.
  Interventions: Behavioral: OACareTools+

INTERVENTIONS:
Behavioral: OACareTools+ — OACareTools+ is a healthcare provider intervention that combines healthcare provider education, customized patient and clinical resources, and technical support from a national organization to facilitate provider counseling on and referral to as well as patient engagement in Walk With Ease. There are 2 main parts to this intervention: 1) Healthcare provider education: The study team will deliver the provider education and resources (including information about Walk With Ease and the established referral process/smartphrase) in a presentation providers at a weekly clinician meeting and in follow-up emails. 2) Implementation: Providers will use the resources to briefly counsel patients about physical activity and Walk With Ease and use the smartphrase to refer patients to Walk With Ease. Patients will register for and participate in the online Walk With Ease program. Patients and providers can seek assistance from the national organization as needed during these processes.
  Other Names: Walk With Ease; Camine Con Gusto

SUMMARY:
The purpose of this pilot study is to test OACareTools+, an intervention for healthcare providers that combines education, patient resources and support from a national organization, to help them make referrals of patients with arthritis to the Walk With Ease program. This intervention was designed to increase referrals of patients with arthritis to the Walk With Ease program.

DETAILED DESCRIPTION:
Participants will be clinicians (n= 50) in a primary care practice and a subset of patients (n=10). The study team will deliver education and resources to providers in a training session about Walk With Ease. After the provider training, providers will use the study resources to refer patients with arthritis to Walk With Ease. Healthcare provider participants will complete surveys after their first referral and at the end of the study (12-months). Patient participants who are referred to Walk With Ease through the OACareTools+ intervention will participate in interviews about their experience (6-weeks) with the referral process. Primary endpoints of the study will be 1) number of healthcare providers that referred patients to Walk With Ease 2) number of Walk With Ease patient participants 3) healthcare provider acceptability and feasibility 4) patient acceptability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare provider participants: currently a healthcare provider or staff person in the UNC pilot clinic
* Patient participants: 18 years or older; received a referral to Walk With Ease from a provider at the UNC pilot clinic; agreed to participate in the phone interview on the post-Walk With Ease evaluation form

Exclusion Criteria:

* Both: non-English speaking

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of healthcare providers who referred patients | 12 months
  Healthcare providers in the pilot clinic who refer patients to the Walk With Ease program using the study referral process and resources
Number of patients who registered for Walk With Ease | 12 months
  Patients from the pilot clinic who are referred to and register in the Walk With Ease program
Healthcare provider acceptability | Measure collected up to 2 months after provider's first referral
  The Acceptability of Intervention Measure is a measure of implementation outcomes, including 4 items ranked on a Likert scale of 1 (completely disagree) to 5 (completely agree), with a summed total ranging from 4-20 where higher scores indicate greater acceptability; measured via electronic survey.
Healthcare provider feasibility | Measure collected up to 2 months after provider's first referral
  The Feasibility of Intervention Measure is a measure of implementation outcomes, including 4 items ranked on a Likert scale of 1 (completely disagree) to 5 (completely agree), with a summed total ranging from 4-20 where higher scores indicate greater feasibility; measured via electronic survey.
Patient acceptability | 6-weeks post- Walk With Ease registration
  The Acceptability of Intervention Measure is a measure of implementation outcomes, including 4 items ranked on a Likert scale of 1 (completely disagree) to 5 (completely agree), with a summed total ranging from 4-20 where higher scores indicate greater acceptability; measured via telephone interview.
Patient usefulness: educational resources | 6-weeks post- Walk With Ease registration
  During a phone interview, patients will be asked, "How helpful were the education materials given to you by your healthcare provider?" They will be asked to use a scale, 0-10, where 0 is not helpful at all and 10 is extremely helpful. Higher scores indicate greater levels of helpfulness.
Patient usefulness: clinician referral to Walk With Ease | 6-weeks post- Walk With Ease registration
  During a phone interview, patients will be asked, "How helpful was it to talk with healthcare provider about physical activity and Walk With Ease?" They will be asked to use a scale, 0-10, where 0 is not helpful at all and 10 is extremely helpful. Higher scores indicate greater levels of helpfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Callahan, PhD, Principal Investigator — UNC Thurston Arthritis Research Center
Locations (1):
- UNC Thurston Arthritis Research Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that support the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC. Data collected include: pre/post walking program assessments, referral count, patient engagement metrics, arthritis outcomes, satisfaction (provider and patient). Qualitative data will be available in the form of a summary.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 and continuing for 36 months following publication. Research study records will be maintained for no less than 6 years following the completion of the study.
Access Criteria: Approved IRB, IEC, or REB and an executed a data use/sharing agreement with UNC.
URL: https://dataverse.unc.edu/